CLINICAL TRIAL: NCT01328821
Title: A Randomized, Double-blind, Placebo-controlled, Single-ascending-dose, Safety, Tolerability, Pharmacokinetics, and Relative Bioavailability Study of CTP-499 in Healthy Adults
Brief Title: Safety, Tolerability, and Pharmacokinetics (PK) of CTP-499
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP505.1001 CTP-499
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Nephropathy
Keywords: Safety; Tolerability; Pharmacokinetics; Healthy volunteers
MeSH Terms: conditions — Diabetic Nephropathies | interventions — 1-(5-hydroxyhexyl)-3,7-dimethylxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Placebo Comparator): Single ascending dose administration of four doses of CTP-499 as tablets under fasting condition.
  8 subjects per dose group will be enrolled with a 3:1 randomization of active drug to placebo.
  Dose levels: 600mg -> 1200mg -> 1800mg -> 2400mg
  Interventions: Drug: CTP-499
- Part B (Active Comparator): Part B will consist of a single 400 mg dose of an immediate release capsule of CTP-499 administered under fasting conditions. In Part B 6 subjects will be enrolled.
  Interventions: Drug: CTP-499

INTERVENTIONS:
Drug: CTP-499 — 600 mg, 1200 mg, 1800 mg and 2400 mg
  Arms: Part A
Drug: CTP-499 — 400 mg immediate release capsule
  Arms: Part B

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of CTP-499 following single dose administration.

DETAILED DESCRIPTION:
This is a double-blind, single ascending dose administration study of four doses of CTP-499. Following dosing safety and tolerability will be assessed. Blood and urine samples will be taken for pharmacokinetics (PK) and bioavailability. Safety assessments will include monitoring of adverse events, vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, 12-lead ECGs, and physical examination findings.

The plasma concentration time data for CTP-499 and its metabolites will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analysis. The primary pharmacokinetics parameters are: Cmax, Tmax, T1/2, AUClast and AUCinf for plasma; relative bioavailability; and Ae and CLr for urine.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* ages 18 to 55 years old
* nonsmokers
* BMI of 18 to 30 kg/m2

Exclusion Criteria:

* Significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders of drug hypersensitivity
* Systolic Blood pressure < 90 or > 140, diastolic bp > 90

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of CTP-499 | 5 days
  Assessments will include monitoring of adverse events, vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, 12 lead ECGs, and physical examination findings. Safety data will be summarized using descriptive statistics for all subjects who receive at least 1 dose. Adverse events will be summarized by frequency. Abnormal laboratory and physical exam findings will be summarized by dose and treatment.

SECONDARY OUTCOMES:
To assess Pharmacokinetics, Pharmacodynamics and relative bioavailability | 2 days
  Pharmacokinetics: individual and mean concentration time profiles will be presented graphically. Alll PK parameters will be summarized by dose group using descriptive statistics (eg n, arithmetic mean, SD, geometric mean, median, CV). Relative bioavailability will be estimated using the geometric mean values of dose normalized AUC for each dose.
  Pharmacodynamics: From the 12 lead ECG data, VR, PR, QRS, QT, QTcF andd QTcB will be reported for each time point and summarized using descriptive statistics. Mean temporal profiles for 12 lead ECG and vital signs will be presented graphically.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tracey, MD, Principal Investigator — Frontage Clinical Services
Locations (1):
- Frontage, Hackensack, New Jersey, United States